CLINICAL TRIAL: NCT07059000
Title: A Phase III, Open-label, Single Arm, Prospective, Multicenter Study to Assess Efficacy and Safety of Kedrion Intravenous Human Normal Immunoglobulin (IVIg) 10% in Adult Patients With Chronic Immune Thrombocytopenia (ITP)
Brief Title: A Study Investigating Intravenous Human Normal Immunoglobulin 10% in Adults With Chronic Immune Thrombocytopenia (ITP)
Acronym: ITP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB072; 2023-507115-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-18; First posted 2025-07-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Primary Immune Thrombocytopenia (ITP)
Keywords: ITP; Primary Immune Thrombocytopenia; Autoimmune Disease; Hemorrhagic Disorders; Hematologic Diseases; Blood Coagulation Disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Autoimmune Diseases; Hemorrhagic Disorders; Hematologic Diseases; Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 2 g/kg Kedrion IVIg 10% (Experimental): Subjects will receive one course of treatment with 2 g/kg of Kedrion IVIg 10% administered over 2 days
  Interventions: Biological: Kedrion IVIG 10%

INTERVENTIONS:
Biological: Kedrion IVIG 10% — (Intravenous) Human Normal Immunoglobulin (IVIg) 10%
  Other Names: KIg 10

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KIg 10 (Intravenous Immunoglobulin 10%) in adult patients with chronic primary ITP

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-70 years of age.
2. Patient and/or legal authorized representative has signed the ICF.
3. Diagnosis of chronic (> 12 months duration) ITP as defined by the International Working Group.
4. Mean screening platelet count of < 30 × 10^9/L from two qualifying counts measured at least one calendar day apart. The first qualifying count can be from historical data if measured within 14 days prior to the first KIg10 infusion. The second qualifying count will be measured within 7 days before the first KIg10 infusion.
5. Platelet count of < 30 × 10^9/L at the Baseline Visit.
6. Patient is willing to comply with all requirements of the protocol.
7. Women of childbearing potential must have a negative urine pregnancy test at screening and agree to employ adequate birth control measures during the study.
8. Authorization to access personal health information.

Exclusion Criteria:

1. Patients with secondary ITP (all forms of immune-mediated thrombocytopenia except primary ITP). e.g., lupus erythematosus, rheumatoid arthritis, drug-related ITP, and Human Immunodeficiency Virus (HIV).
2. Patients with Evans Syndrome.
3. Patients known to be infected with hepatitis B virus, hepatitis C virus, or HIV.
4. History of thrombotic events including deep vein thrombosis, cerebrovascular accident, pulmonary embolism, transient ischemic attacks, or myocardial infarction.
5. Patient with a history of hypersensitivity to IVIg, other injectable forms of IVIg, or to any of the excipients.
6. Patient unresponsive previously to IVIg or anti-D Ig treatment.
7. Patient with known Immunoglobulin A (IgA) deficiency and antibodies against IgA.
8. Splenectomy within 4 weeks of the Baseline Visit or planned splenectomy throughout the study period.
9. Subjects with known inherited thrombocytopenia. e.g., MYH-9 disorders.
10. Subjects with myelodysplastic syndrome (MDS).
11. Administration of IVIg, anti-D immunoglobulin, mercaptopurine, vinca alkaloid, or platelet enhancing drugs (including thrombopoietin receptor agonists [TPO-RA], immunosuppressive, or other immunomodulatory drugs) within 3 weeks of the Baseline Visit, except for:

    1. patients on a stable dose of TPO-RA within 4 weeks of the Baseline Visit
    2. patients on a stable dose of Mycophenolate Mofetil within 3 months of the Baseline Visit
    3. patients on stable dose of Danazol within 3 months of the Baseline Visit
    4. long-term corticosteroid therapy for ITP, when the dose had been stable within 3 weeks of the Baseline Visit and no dosage change was planned until the EOS Visit
    5. long-term azathioprine cyclophosphamide or attenuated androgen therapy when the dose had been stable within 3 months of the Baseline Visit, and no dosage change was planned until after study completion.
12. Received any blood, blood product, or blood derivative within 1 month of the Baseline Visit.
13. Received rituximab within 6 months of the Baseline Visit.
14. Had a platelet transfusion or receipt of blood products containing platelets within 7 days of Visit 1 (Day 1).
15. Received recombinant activated factor VII within 7 days of the Baseline Visit.
16. Had therapy with live attenuated virus vaccines within 3 months of the Baseline Visit.
17. Use of loop diuretics within 1 week of the Baseline Visit.
18. Patients at high risk of thrombotic events.
19. Uncontrolled hypertension [i.e., diastolic blood pressure >100 mmHg and/or systolic blood pressure >160 mmHg]. If a single measure exceeds this limit, a triple repeat measurement may be performed and the average of the three measurements used.
20. Congestive heart failure as per New York Heart Association III/IV, cardiomyopathy, cardiac arrhythmia associated with thromboembolic events (e.g., atrial fibrillation), unstable or advanced ischemic heart disease, hyperviscosity.
21. Patients with significant protein losing enteropathy, nephrotic syndrome, or lymphangiectasia.
22. Patients with hyperproteinemia, increased serum viscosity, and/or hyponatremia.
23. Severe liver or kidney disease (normal reference ranges of laboratory doing the analysis):

    1. alanine aminotransferase (ALT) or aspartate amino transferase (AST) 2.5x > upper limit of normal
    2. creatinine > 120 μmol/L
    3. blood urea nitrogen (BUN) > 2.5x the upper limit of normal.
24. Signs of severe anemia: Hemoglobin of less than 7 g/dL, hemodynamically unstable due to active bleeding, and/or when evidence of end-organ ischemia secondary to severe anemia is present.
25. Body mass index > 40 kg/m2 or an IVIg dose that puts the patient at risk of fluid overload.
26. History of a malignant disease within 3 years of the Baseline Visit other than properly treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin.
27. Patient has participated in an interventional, investigational clinical study within 30 days of the Baseline Visit.
28. Any condition that the Investigator believes is likely to interfere with evaluation of the study drug or with satisfactory conduct of the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects with response (R) | Treatment to day 14
  Assess the responder rate by measuring the platelet count increase according to the Response (R) definition and the absence of bleeding during the evaluation period

SECONDARY OUTCOMES:
Number and rate of subjects with complete response (CR) | Treatment to day 14
  Assess the clinical response rate by measuring the platelet count increase and absence of bleeding according to the Complete Response (CR)
Time to platelet count response | Treatment to day 14
  Assess the time from starting treatment to time of achievement of CR or R
Duration of response | 14 days after treatment to end of study
  Measured from achievement of CR or R to loss of CR or R
Regression of hemorrhages | Day 1 (Visit 1) to Day 30 (End of Study Visit)
  Time to stop bleedings
Platelet count assessment | Day 1 (Visit 1) to Day 30 (End of Study Visit)
  Assess the maximum platelet count and time to achieve the maximum platelet count
Assess safety and tolerability | Day 1 (Visit 1) to Day 30 (End of Study Visit)
  Number and percentage of all adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Calcinai, MD, Study Director — Kedrion S.p.A.
Locations (27):
- United States (2):
  - University of Southern California, Los Angeles, California
  - East Carolina University, Greenville, North Carolina
- Czechia (2):
  - Vseobecna Fakultni Nemocnice v Praze, Prague, Prague
  - Fakultni Nemocnice Brno, Brno, South Moravian
- Germany (2):
  - Onkologisches Zentrum Donauwörth Neudegger - Onkomedeor Onkologische Zentren, Donauwörth, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
- Italy (5):
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara, Novara
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste, Trieste
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino, Turin
  - AULSS 8 Berica - Ospedale San Bortolo Di Vicenza, Vicenza, Vicenza
- Romania (3):
  - Coltea - Spital Clinic, Bucharest, București
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca, Cluj
  - Spitalul Filantropia - Craiova, Craiova, Dolj
- Serbia (2):
  - Univerzitetski Klinicki Centar Srbije, Belgrade
  - Klinicko-Bolnicki Centar Zemun, Belgrade
- Spain (4):
  - Complejo Asistencial Universitario de Burgos - Hospital Universitario de Burgos, Burgos, Burgos
  - Instituto De Investigacion Biomedica De A Coruna - Virologia Clinica, A Coruña, La Coruña
  - Complejo Hospitalario Ruber Juan Bravo, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
- Turkey (Türkiye) (7):
  - Ankara Üniversitesi Tip Fakültesi - Cebeci Arastirma ve Uygulama Hastanesi, Ankara, Ankara
  - Kocaeli Üniversitesi Arastirma ve Uygulama Hastanesi, Ankara, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Yenimahalle, Ankara
  - Trakya Üniversitesi Saglik Arastirma ve Uygulama Merkezi, Edirne, Edirne
  - Ege Universitesi Tip Fakultesi, Izmir, İzmir
  - VM Medical Park Mersin Hastanesi, Mersin, Mersin
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi, Adapazarı, Sakarya

IPD SHARING:
Plan to Share IPD: No
Publishing of data and IPD that underlie results in the publication will be determined at study completion to comply with ICJME minimum requirements.